CLINICAL TRIAL: NCT05539066
Title: Application of AI Health Assistant in Out of Hospital Management of Patients With Type 2 Diabetes
Brief Title: AI Health Assistant and Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liping Gu, Deputy chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21Y11904800
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Health Behavior; Type2 Diabetes Mellitus
Keywords: Type 2 Diabetes; AI health assistant; Off hospital management
MeSH Terms: conditions — Health Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI health assistant (Experimental): An AI health assistant suitable for diabetes patients has been developed. It has the functions of automatically uploading blood pressure, blood glucose data, intelligent reminder, automatic analysis of reports inside and outside the hospital, intelligent question and answer, etc. it is simple to operate, highly interactive, and maximizes the management level of diabetes patients outside the hospital.
  Interventions: Device: AI health assistant
- Routine treatment group (No Intervention): Perform routine management and follow-up without using AI health assistant

INTERVENTIONS:
Device: AI health assistant — To study the advantages of AI health assistant management group compared with conventional management group in terms of comprehensive compliance rate, metabolic index level, hypoglycemia incidence rate, and mastery of diabetes related knowledge.
  Arms: AI health assistant

SUMMARY:
The developed health assistant has the functions of intelligent analysis of health data inside and outside the hospital, health reminder, etc. The advantages of AI health assistant management group compared with conventional management group in terms of comprehensive compliance rate, metabolic index level, hypoglycemia incidence rate was further studied.

DETAILED DESCRIPTION:
1. The investigators have developed an AI health assistant suitable for diabetes patients, which has the functions of automatically uploading blood pressure, blood glucose data, intelligent reminder, automatic analysis of reports inside and outside the hospital, intelligent question and answer, etc. it is simple to operate, highly interactive, and maximizes the management level of diabetes patients outside the hospital.
2. Through AI personal health assistant, 196 diabetes patients were managed to further improving the comprehensive compliance rate of metabolic indicators such as blood glucose and blood pressure of diabetes patients, improving the patients' self-management ability.

ELIGIBILITY:
Inclusion Criteria:

The diagnostic criteria of T2DM patients are the diagnostic criteria of the 2017 China guidelines for the prevention and treatment of type 2 diabetes HbA1c 7.5-13% Age: 18-65y BMI 18.5-30kg/m2 The course of disease is less than 5 years Have good cognitive ability and can correctly use health assistants

Exclusion Criteria:

Acute complications of diabetes (diabetes ketosis, etc.) Diabetes complicating pregnancy or preparing for pregnancy HbA1c < 7.5% or > 13% Age < 18y or age > 65y Pre pregnancy BMI < 18.5 or > 30kg / m2 Severe liver and kidney dysfunction (ALT greater than 2.5 times the upper limit of normal, EGFR less than 45 ml / min / 1.73m2) Using drugs that may affect blood glucose are being used (including steroids, hydroxyprogesterone hexanoate, anti AIDS drugs, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c compliance rate | 6 months
  Compliance rate of HbA1c < 7%
Blood pressure compliance rate | 6 months
  Proportion of patients with blood pressure < 130 / 80mmHg
Compliance rate of total cholesterol | 6 months
  Proportion of patients with total cholesterol < 4.5mmol/l
Compliance rate of BMI (Body Mass Index) | 6 months
  Proportion of patients with BMI < 24 kg/m2

SECONDARY OUTCOMES:
Incidence of hypoglycemia | 6 months
  Number of attacks with blood glucose less than 3.8mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Yufan Wang, doctor, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No